CLINICAL TRIAL: NCT01667315
Title: Minimum Effective Volume of 0.375% Bupivacaine in Ultrasound- and Nerve Stimulator-guided Interscalene Brachial Plexus Block for Shoulder Surgery
Brief Title: Minimum Effective Volume of 0.375% Bupivacaine in Interscalene Brachial Plexus Block
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Fernando Saldanha de Almeida, Principal Investigator, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Bupivacaine 0,375%
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Shoulder Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine (Experimental): Bupivacaine 0,375%
  Interventions: Drug: Bupivacaine 0,375%

INTERVENTIONS:
Drug: Bupivacaine 0,375% — Positive or negative block results in a 1-mL reduction or increase in volume, respectively.

SUMMARY:
The use of ultrasound in regional anesthesia enables reduction in the local anesthetic volume. The present study aimed to determine the minimum effective volume of 0.375% bupivacaine with epinephrine for interscalene brachial plexus block for shoulder surgery. Following approval by the Research Ethics Committee, patients with a physical condition of I or II according to the American Society of Anesthesiologists, between 21 and 65 years old and subjected to elective surgery of the shoulder and interscalene brachial plexus block will be recruited. The volume of the anesthetic will be determined using a step-up/step-down method and based on the outcome of the preceding block. Positive or negative block results in a 1mL reduction or increase in volume, respectively. The success of the block is defined as the presence of motor block in two muscle groups and the absence of thermal and pain sensations in the necessary dermatomes within 30 minutes of the injection. Diaphragmatic paralysis, pulmonary function and analgesia will be quantified at 30 minutes, 4 and 6 hours. Data will undergo statistical analysis in order to determine minimum effective volume of 0.375% bupivacaine and, secondarily, the maximum volume that maintains the diaphragmatic function, evaluate diaphragm paralysis and its influence in pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years
* Candidates for an elective surgical intervention on the shoulder with indication for anesthesia via brachial plexus block
* Physical condition of I or II according to the American Society of Anesthesiologists
* Body mass index up to 35 kg.m-2

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Cognitive impairment or active psychiatric condition
* Infection at the site of the puncture for the block
* Coagulopathy
* Bupivacaine allergy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Minimum effective volume of 0,375% bupivacaine | 30 minutes
  Minimum effective volume of 0,375% bupivacaine with epinephrine in ultrasound-guided interscalene brachial plexus block for shoulder surgery

SECONDARY OUTCOMES:
Maximum 0,375% bupivacaine volume that maintains the diaphragmatic function | Before block, 10, 20 and 30 minutes, 4 and 6 hours after
  Maximum effective volume of 0,375% bupivacaine with epinephrine in ultrasound-guided interscalene brachial plexus block for shoulder surgery without diaphragmatic block
Pulmonary function | Before block, 30 minutes, 4 and 6 hours after
  Spirometric evaluation of forced vital capacity
Diaphragmatic Function | Before block, 30 minutes, 4 and 6 hours after
  Diaphragmatic movement on ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil